CLINICAL TRIAL: NCT01542619
Title: A Randomized, Placebo-controlled, Single Center, 5 Cohort Dose Escalation Trial to Investigate Safety and Pharmacokinetics of rVIIa-FP (CSL689) in Comparison to Placebo in Healthy Male Human Volunteers
Brief Title: A Safety and Pharmacokinetics Study of a Recombinant Fusion Protein Linking Coagulation Factor VIIa With Albumin (rVIIa-FP) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL689_1001; 2011-004568-32 (EudraCT Number)
Record Dates: First submitted 2012-02-26; First posted 2012-03-02 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2013-03

CONDITIONS: Healthy
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- rVIIa-FP (Experimental)
  Interventions: Biological: rVIIa-FP
- Placebo (0.9% normal saline) (Placebo Comparator)
  Interventions: Biological: Placebo (0.9% normal saline)

INTERVENTIONS:
Biological: rVIIa-FP — Recombinant VIIa-FP (rVIIa-FP) is a fusion protein linking coagulation factor VIIa with albumin and will be administered by intravenous infusion in escalating doses up to 1000 mcg/kg. Participants will receive pre-treatment with an oral anticoagulant starting 7 days prior to administration of study product and continuing for 7 days after study product has been administered.
  Arms: rVIIa-FP
Biological: Placebo (0.9% normal saline) — Placebo will be administered by intravenous infusion. Participants will receive pre-treatment with an oral anticoagulant starting 7 days prior to administration of placebo and continuing for 7 days after placebo has been administered.
  Arms: Placebo (0.9% normal saline)

SUMMARY:
This is a first in man, prospective, single-center, randomized, double-blind, dose-escalation cohort study to investigate tolerability, safety and pharmacokinetics of rVIIa-FP in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 18 and 35 years of age, both inclusive.
* Body weight between 50.0 and 100.0 kg, both inclusive.
* Body mass index (BMI) between 18.0 and 29.9 kg/m2, both inclusive.
* Written informed consent for study participation obtained before undergoing any study specific procedures.

Exclusion Criteria:

* Subjects at increased cardiovascular risk.
* Any clinical sign or known history of atherosclerosis or thromboembolic events.
* A subject considered at high risk of thromboembolic events confirmed either from history or by thrombophilia screening test.
* Subjects with significant elevation of cholesterol level.
* Renal dysfunction.
* Overt bleeding.
* Smokers with positive cotinine test at screening.
* Participation in any other trial investigating a procoagulant within the last six months prior to screening.
* Known or suspected hypersensitivity to the investigational medicinal product (IMP), or to any excipients of the IMP.
* Contraindications to Warfarin (Coumadin®).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The frequency of related Adverse Events (AEs) to rVIIa-FP. | 28 days
Number of subjects who develop inhibitors against Factor VII (FVII). | 28 days
Number of subjects who develop antibodies against rVIIa-FP. | 28 days

SECONDARY OUTCOMES:
Area under curve to the last sample with quantifiable drug concentration (AUC0-t) of a single dose of rVIIa-FP | 120 hours
Half- life (t1/2) of a single dose of rVIIa-FP | 120 hours
Incremental recovery (IR) of rVIIa-FP | 120 hours
Clearance (Cl) of a single dose of rVIIa-FP | 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alex Veldman, M.D., Study Director — CSL Behring
Locations (1):
- Phase I Unit, Berlin, Germany

REFERENCES:
- [Result] Golor G, Bensen-Kennedy D, Haffner S, Easton R, Jung K, Moises T, Lawo JP, Joch C, Veldman A. Safety and pharmacokinetics of a recombinant fusion protein linking coagulation factor VIIa with albumin in healthy volunteers. J Thromb Haemost. 2013 Nov;11(11):1977-85. doi: 10.1111/jth.12409. PMID 24112951